CLINICAL TRIAL: NCT04108624
Title: A Multimodality Approach to Minimal Residual Disease Detection to Guide Post-Transplant Maintenance Therapy in Multiple Myeloma (MRD2STOP)
Brief Title: Study to Assess for Measurable Residual Disease (MRD) in Multiple Myeloma Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB19-0339
Record Dates: First submitted 2019-09-19; First posted 2019-09-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MRD2STOP ARM (Experimental)
  Interventions: Other: Screening Phase; Device: Discontinuation Phase

INTERVENTIONS:
Other: Screening Phase — This will identify subjects who are MRD (minimal residual disease) negative and eligible for the discontinuation phase.
Device: Discontinuation Phase — Patients will undergo discontinuation of their maintenance therapy if they are MRD negative by PET/CT (Positron Emission Tomography/Computed Tomography), flow cytometry and next generation sequencing

SUMMARY:
This study is to assess for Measurable Residual Disease (MRD) in multiple myeloma at a deeper level than what is currently available by combining novel imaging and laboratory techniques, determine if patients who are MRD-negative by these multiple modalities can safely and effectively discontinue post-transplant maintenance therapy, and determine if liquid biopsies is a more accurate and/or less invasive sampling technique for multiple myeloma.

The purpose of this research is to determine if patients who are MRD-negative by multiple modalities ("multimodality MRD-negative") can safely and effectively discontinue post-transplant maintenance therapy (single agent lenalidomide, pomalidomide, bortezomib, or ixazomib) after receiving at least one year of maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females > 18 years of age
* ECOG performance status less than or equal to 2 (Karnofsky > 60%)
* Patients with a diagnosis of multiple myeloma who have undergone initial treatment, with or without autologous stem cell transplant, and currently treated with single-agent maintenance therapy (lenalidomide, pomalidomide, bortezomib, daratumumab, or ixazomib) for a duration of at least 1 year. The 1 year duration can include time spent receiving at least 8 cycles of doublet or triplet induction regimens OR multi-agent post-transplant maintenance prior to conversion to single agent maintenance therapy.
* Patients must have had their most recent bone marrow testing within the last 2 years and negative for MRD by flow cytometry (with a sensitivity of at least 10-5) or by NGS with a sensitivity of at least 10-5.
* Patients must have achieved a CR (CR) by IMWG consensus response criteria. For patients with a persistent low level paraprotein ('M-spike'), mass spectrometry may be used to determine if the paraprotein is significant or not. Results of mass spectrometry may be used to supercede results of serum protein electrophoresis.
* Patients must have a most recent PET/CT within the last 1.5 years without evidence of myeloma disease.
* Must have baseline bone marrow sample that can be used for clonality identification for NGS and mass spectrometry if not already performed.
* Willing and able to undergo a bone marrow biopsy and aspiration.
* Ability to understand and the willingness to sign a written informed consent document.
* Females of childbearing potential (FCBP) must agree to use 2 reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) if continued on lenalidomide as part of standard of care and 2) for at least 28 days after discontinuation of lenalidomide
* All participants in the US must have already been consented to and registered into the mandatory Revlimid REMS® program and be willing and able to comply with the requirements of Revlimid REMS®.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the intervention are eligible for this trial.

Exclusion Criteria:

* Progressive disease as determined per IMWG consensus response criteria.
* Have not met the criteria for CR by IMWG consensus response criteria.
* MRD-positive disease by flow cytometry, NGS (1 in 1,000,000 cells), or PCR.
* Concomitant hematologic malignancy.
* Known or suspected amyloidosis.
* Unwilling to undergo a bone marrow biopsy.
* Unwilling to discontinue maintenance therapy.
* Any clinically significant medical disease or condition that, in the Treating Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Determine the MRD conversion rate | 3 years
  Determine the MRD conversion rate from 1 in 1,000,000 cells and 1 in 10,000,000 cells negative to positive after discontinuation of maintenance therapy.
Median Progression Free Survival rate | 3 years
  Assess progression free survival of double MRD-negative (1 in 1,000,000 cells negative/1 in 10,000,000 cells negative) patients and of the 1 in 1,000,000 cells negative/1 in 10,000,000 cells positive patients who have discontinued maintenance therapy
Median overall survival rate | 3 years
  Assess overall survival of double MRD-negative (1 in 1,000,000 cells negative/1 in 10,000,000 cells negative) patients and of the 1 in 1,000,000 cells negative/1 in 10,000,000 cells positive patients who have discontinued maintenance therapy.

SECONDARY OUTCOMES:
NGS-based Minimal Residual Disease testing determined by the ClonoSeq assay | 3 years
  Determine the feasibility of performing NGS-based MRD testing of bone marrow aspirate samples that have undergone CD138+ immunomagnetic cell separation (i.e. 1 in 10,000,000 cells depth) will be determined by the rate of achieving 20 million cells in raw aspirate sample with a sufficient DNA for analysis as determined by the ClonoSeq assay.
Determine the difference in MRD detection by NGS | 3 years
  Determine the difference in MRD detection by NGS in the bone marrow at depths of 1 in 1,000,000 cells and 1 in 10,000,000 cells.

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Jakubowiak, MD, Principal Investigator — University of Chicago
Locations (1):
- University Of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States